CLINICAL TRIAL: NCT06906692
Title: Evaluation of Antibody Titles After Meningococcal Vaccination in Patients With Myasthenia Gravis and Neuromyelitis Optica Candidate to Complement Inhibitors Therapy
Brief Title: Meningococcal Vaccination in Patients on Complement Inhibitors
Acronym: Vax_MenACWY
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7355
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Myasthenia Gravis Generalised; Vaccination; Complement System; Neuromyelitis Optica Spectrum Disease (NMOSD)
MeSH Terms: interventions — Serum Bactericidal Antibody Assay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum Bactericidal Assay — The Serum Bactericidal Assay (SBA) will be used for the analysis of the antibody titer, which represents a valid surrogate for the efficacy of the tetravalent vaccine. Subjects' sera will be serially diluted and incubated with a solution containing a certain strain of meningococcus. At this point, an exogenous source of rabbit complement will be added. Bactericidal activity will be assessed against controls. Neutralizing antibody titers will be defined as the highest dilution of sera at which at least 50% of bacteria death occurs. Antibody titers will be considered protective with a cut-off greater than or equal to 1:8.

SUMMARY:
Myasthenia gravis is an autoimmune neurological disorder caused by autoantibodies directed predominantly against components of the postsynaptic membrane of the neuromuscular junction. Anti-aquaporin-4 antibody-associated neuromyelitis optica (AQP4-IgG) is an autoimmune inflammatory disease of the central nervous system (CNS) characterized by three main clinical manifestations: transverse myelitis, optic neuritis, and postrema area syndrome. Over the past five years, the FDA and EMA have approved complement inhibitor drugs for the treatment of generalized myasthenia gravis with anti-AChR antibody positivity and for neuromyelitis optica spectrum disorders with anti-AQP4 antibody positivity. Eculizumab is a humanized monoclonal antibody that binds to the C5 fragment of the human complement specifically and with high affinity, inhibiting its cleavage in C5a and C5b and preventing the formation of the membrane attachment C5b-9 complex (MAC) of the terminal portion of the complement cascade. This monoclonal antibody maintains the early components of complement activation (C3b), which are essential for the opsonization of microorganisms and the clearance of immune complexes. Ravulizumab is a monoclonal antibody derived from eculizumab, through the substitution of four specific amino acids, which binds specifically to complement protein C5. These substitutions increase the dissociation of the monoclonal antibody from the C5 fragment within the endosome and promote the recycling of the neonatal Fc receptor-mediated unbound antibody, extending its half-life and duration of action up to an interval of 8 weeks. Zilucoplan is a synthetic macrocyclic peptide composed of 15 amino acids that specifically binds the complement protein C5, inhibiting its cleavage into C5a and C5b by C5 convertase, which results in an underregulation of MAC assembly and cytolytic activity. In addition, this drug binds the C5b fraction of C5, creating a steric encumbrance for the binding of C5b to C6 and preventing subsequent assembly of the MAC if any C5b is formed. Due to their mechanism of action, eculizumab, ravulizumab and zilucoplan result in an increased susceptibility of the patient to systemic infections by encapsulated bacteria (S. pneumoniae, H. influenzae, N. meningitidis). To reduce the risk of infection, all patients should be vaccinated against serogroups A, B, C, W, Y at least 2 weeks prior to treatment; patients who start treatment before 2 weeks after administration of meningococcal vaccines should be given appropriate antibiotic prophylaxis for up to 2 weeks after vaccination. Currently, there is no global agreement on the vaccination schedule to be followed after the first dose. According to Italian guidelines, a booster dose is recommended for the monovalent vaccine only at least 1 month after the first administration and a period of antibiotic prophylaxis beyond the first two weeks after the first doses is not indicated. The primary objective of the study is to evaluate the antibody titles after tetravalent meningococcal vaccination (serogroups A, C, W, Y) in patients candidate to complement inhibitors therapy.

ELIGIBILITY:
Inclusion Criteria:

* Study Participant must be ≥ 18 years old;
* Diagnosis of anti-AChR positive generalized Myasthenia Gravis or Positive anti-AQP4 NMOSD;
* Need for therapy with complement inhibitor drugs according to the therapeutic indications approved by AIFA;
* Possibility of follow-up in the reference centre;
* Signing of the Informed Consent to the Study.

Exclusion Criteria:

* Age < 18 years;
* Poor Compliance with Drug Therapy
* Insufficient availability of Clinical Information;
* Current Neoplasm or Infection at the Time of Collection of Biological Samples;
* Refusal to Sign the Informed Consent to the Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with generalized myasthenia gravis positive for anti-AChR antibodies and neuromyelitis optica spectrum disorder positive for anti-AQP4 antibodies, candidates for treatment with complement inhibitor drugs, belonging to the IRCCS Fondazione Policlinico A. Gemelli on an outpatient basis, who meet the inclusion and exclusion criteria of the study, will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of antibody titres after tetravalent meningococcal vaccine (serogroups A, C, W, Y) in patients candidate to complement inhibitors therapy | 24 months
  Antibody titers will be considered protective with a cut-off greater than or equal to 1:8. The primary endpoint of this study is to evaluate the number of patients that will develope a protective titer of neutralizing antibodies against meningococcus A, C, W, Y after vaccination

SECONDARY OUTCOMES:
Evaluation of chronic intake of immunosuppressive therapies | 24 months
  Evaluation of correlations between antibody titles and chronic intake of immunosuppressive therapies

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Iorio, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico A. Gemelli IRCCS, Rome, RM, Italy